CLINICAL TRIAL: NCT01154088
Title: Immunogenicity and Safety Study of One Dose of GSK Biologicals' Meningococcal Vaccine GSK 134612 (Blinded Lots) Versus One Dose of Mencevax™ ACWY in Healthy Subjects Aged 18-25 Years
Brief Title: Immunogenicity and Safety of Meningococcal Vaccine GSK 134612 Versus Mencevax™ ACWY in Healthy 18-25 Year Olds
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 114248
Record Dates: First submitted 2010-06-29; First posted 2010-06-30 (Estimated); Results first posted 2018-11-26 (Actual); Last update posted 2018-11-26 (Actual); Status verified 2018-05

CONDITIONS: Infections, Meningococcal
Keywords: Adolescent; Vaccine, conjugate; Adult; Neisseria meningitidis; Immunogenicity; Meningococcal vaccine; Safety
MeSH Terms: conditions — Meningococcal Infections | interventions — PsACWY vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (3):
- Group A (Experimental)
  Interventions: Biological: GSK Biologicals' meningococcal serogroup A, C, W-135, Y tetanus toxoid conjugate investigational vaccine [GSK 134612]
- Group B (Experimental)
  Interventions: Biological: GSK Biologicals' meningococcal serogroup A, C, W-135, Y tetanus toxoid conjugate investigational vaccine [GSK 134612]
- Group C (Active Comparator)
  Interventions: Biological: Mencevax ACWY

INTERVENTIONS:
Biological: Mencevax ACWY — One dose, Subcutaneous injection
  Arms: Group C
Biological: GSK Biologicals' meningococcal serogroup A, C, W-135, Y tetanus toxoid conjugate investigational vaccine [GSK 134612] — One dose, Intramuscular injection
  Arms: Group A; Group B

SUMMARY:
The purpose of the observer-blinded study is to determine the immunogenicity and safety of one dose of GlaxoSmithKline (GSK) Biologicals' meningococcal vaccine GSK 134612 compared to one dose of Mencevax™ ACWY in healthy subjects 18-25 years of age. In addition, this study will compare the immunogenicity of two lots of GSK's 134612 vaccine.

ELIGIBILITY:
Inclusion Criteria:

All subjects must satisfy all of the following criteria at study entry:

* Subjects whom the investigator believes they can and will comply with the requirements of the protocol will be enrolled in the study.
* A male or female between, and including, 18 and 25 years of age the time of the vaccination.
* Written informed consent obtained from the subject.
* Healthy subjects as established by medical history and clinical examination before entering into the study.
* Female subjects of non-childbearing potential may be enrolled in the study.
* Female subjects of childbearing potential may be enrolled in the study, if the subject:

  * has practiced adequate contraception for 30 days prior to vaccination, and
  * has a negative pregnancy test on the day of vaccination, and
  * has agreed to continue adequate contraception during the entire treatment period and for 2 months after vaccination.

Exclusion Criteria:

The following criteria should be checked at the time of study entry. If any exclusion criterion applies, the subject must not be included in the study:

* Use of any investigational or non-registered product other than the study vaccine(s) within 30 days preceding the dose of study vaccine, or planned use during the study period.
* Chronic administration of immunosuppressants or other immune-modifying drugs within six months prior to vaccination. (For corticosteroids, this will mean prednisone <10 mg/day, or equivalent, is allowed. Inhaled and topical steroids are allowed).
* Planned administration/administration of a vaccine not foreseen by the study protocol within one month of the dose of vaccine, with the exception of any licensed inactivated influenza vaccine, including H1N1 vaccine.
* Previous vaccination with meningococcal polysaccharide vaccine within the last five years.
* Previous vaccination with meningococcal conjugate vaccine.
* Previous vaccination with tetanus-toxoid or tetanus-toxoid containing vaccine within the last month.
* History of meningococcal disease.
* Seropositive for HIV or HBsAg (for subjects in the Philippines only).
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus infection, based on medical history and physical examination.
* A family history of congenital or hereditary immunodeficiency, until the immune competence of the potential vaccine recipient has been demonstrated.
* History of reactions or allergic disease likely to be exacerbated by any component of either vaccine.
* History of any neurologic disorders, including Guillain-Barré Syndrome.
* Major congenital defects or serious chronic illness.
* Acute disease at the time of enrolment.
* Administration of immunoglobulins and/or any blood products within the three months preceding the dose of study vaccine or planned administration during the study period.
* Pregnant or lactating female.
* History of chronic alcohol consumption and/or drug abuse.
* Female planning to become pregnant or planning to discontinue contraceptive precautions.
* Bleeding disorders, such as thrombocytopenia, or subjects on anti-coagulant therapy.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1170 (Actual)
Dates: Start 2010-08-27; Primary Completion 2010-12-30 (Actual); Study Completion 2010-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- GSK Investigational Site, Panama City, Panama
- GSK Investigational Site, City of Muntinlupa, Philippines
- GSK Investigational Site, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Lupisan S, Limkittikul K, Sosa N, Chanthavanich P, Bianco V, Baine Y, Van der Wielen M, Miller JM. Meningococcal polysaccharide A O-acetylation levels do not impact the immunogenicity of the quadrivalent meningococcal tetanus toxoid conjugate vaccine: results from a randomized, controlled phase III study of healthy adults aged 18 to 25 years. Clin Vaccine Immunol. 2013 Oct;20(10):1499-507. doi: 10.1128/CVI.00162-13. Epub 2013 Jul 24. PMID 23885033
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 114248 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 114248 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 114248 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 114248 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 114248 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 114248 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Groups:
- Nimenrix-A Group: Healthy male and female subjects, aged 18-25 years, received a single dose of Nimenrix Lot A vaccine administered by intramuscular injection in the deltoid region of the non-dominant arm.
- Nimenrix-B Group: Healthy male and female subjects, aged 18-25 years, received a single dose of Nimenrix Lot B vaccine administered by intramuscular injection in the deltoid region of the non-dominant arm.
- Mencevax Group: Healthy male and female subjects, aged 18-25 years, received a single dose of Mencevax vaccine administered by subcutaneous injection in the upper region of the non-dominant arm.
Period: Overall Study
Arm/Group | Nimenrix-A Group | Nimenrix-B Group | Mencevax Group
Started | 390 | 390 | 390
Completed | 386 | 384 | 383
Not Completed | 4 | 6 | 7
Not completed — Lost to Follow-up | 4 | 6 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nimenrix-A Group | Nimenrix-B Group | Mencevax Group | Total
Number analyzed (Participants) | 390 | 390 | 390 | 1170
Age, Continuous [Mean (Standard Deviation); unit: Years] | 20.8 (2.14) | 20.9 (2.10) | 20.6 (1.94) | 20.77 (2.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 197 | 225 | 204 | 626
  Male | 193 | 165 | 186 | 544
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African heritage/African American | 16 | 13 | 17 | 46
  Asian - Central/South Asian heritage | 0 | 1 | 0 | 1
  Asian - East Asian heritage | 2 | 1 | 2 | 5
  Asian - Japanese heritage | 0 | 0 | 1 | 1
  Asian - South East Asian heritage | 258 | 259 | 257 | 774
  White - Arabic/North African heritage | 1 | 0 | 0 | 1
  White - Caucasian/European heritage | 13 | 14 | 13 | 40
  Other | 100 | 102 | 100 | 302

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Vaccine Response for Serum Bactericidal Assay Using Rabbit Complement Against Neisseria Meningitides Serogroups A, C, W-135, Y (rSBA-MenA, rSBA-MenC, rSBA-MenW-135 and rSBA-MenY) Antibodies
Description: Vaccine response defined as: for initially seronegative subjects, antibody titer greater than or equal to (≥) 1:32 and for initially seropositive subjects: antibody titer ≥ 4 fold the pre-vaccination antibody titer. The analysis was performed with the GSK rSBA assay.
Time Frame: At Month 1
Population: The analysis was performed on the According-To-Protocol (ATP) cohort for immunogenicity, which included all evaluable subjects for whom immunogenicity measures were available. This primary outcome and the statistical analyses performed for this outcome concern the Nimenrix-A Group and Mencevax Group only.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix-A Group | Nimenrix-B Group | Mencevax Group
Number analyzed (Participants) | 358 | 353 | 357
Participants
  rSBA-MenA: number analyzed (Participants) | 302 | 298 | 293
  rSBA-MenA | 239 | 238 | 216
  rSBA-MenC: number analyzed (Participants) | 346 | 342 | 353
  rSBA-MenC | 324 | 327 | 332
  rSBA-MenW-135: number analyzed (Participants) | 338 | 327 | 337
  rSBA-MenW-135 | 328 | 312 | 304
  rSBA-MenY | 334 | 324 | 308
Statistical Analysis 1: Comparison: Nimenrix-A Group vs Mencevax Group; Demonstration of the non-inferiority of the vaccine response induced by Nimenrix conjugate vaccine (Nimenrix Lot A) when compared to the licensed Mencevax for Neisseria meningitidis (N. meningitidis) serogroups A as measured by serum bactericidal antibodies using baby rabbit complement (rSBA) at GSK; Test type: Non-Inferiority — Criterion for non-inferiority: For each serogroup separately, the lower limit (LL) of the 2-sided standardised asymptotic 95% confidence interval (CI) for the group difference (Nimenrix-A Group minus Mencevax Group) in the percentage of subjects with bactericidal vaccine response would be greater than or equal to (≥) the pre-defined clinical limit of -10%; Difference in vaccine response rate = 5.42, 95% CI 2-sided [-1.41 to 12.25]
Statistical Analysis 2: Comparison: Nimenrix-A Group vs Mencevax Group; Demonstration of the non-inferiority of the vaccine response induced by Nimenrix conjugate vaccine (Nimenrix Lot A) when compared to the licensed Mencevax for Neisseria meningitidis (N. meningitidis) serogroups C as measured by serum bactericidal antibodies using baby rabbit complement (rSBA) at GSK; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Difference in vaccine response rate = -0.41, 95% CI 2-sided [-4.11 to 3.25]
Statistical Analysis 3: Comparison: Nimenrix-A Group vs Mencevax Group; Demonstration of the non-inferiority of the vaccine response induced by Nimenrix conjugate vaccine (Nimenrix Lot A) when compared to the licensed Mencevax for Neisseria meningitidis (N. meningitidis) serogroups W-135 as measured by serum bactericidal antibodies using baby rabbit complement (rSBA) at GSK; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Difference in vaccine response rate = 6.83, 95% CI 2-sided [3.28 to 10.78]
Statistical Analysis 4: Comparison: Nimenrix-A Group vs Mencevax Group; Demonstration of the non-inferiority of the vaccine response induced by Nimenrix conjugate vaccine (Nimenrix Lot A) when compared to the licensed Mencevax for Neisseria meningitidis (N. meningitidis) serogroups Y as measured by serum bactericidal antibodies using baby rabbit complement (rSBA) at GSK; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Difference in vaccine response rate = 7.02, 95% CI 2-sided [2.63 to 11.58]

2. Primary Outcome: rSBA-MenA, rSBA-MenC, rSBA-MenW-135 and rSBA-MenY Titers
Description: Titers are presented as geometric mean titers (GMTs). All subjects underwent testing with the GSK rSBA assay for all 4 serogroups.
Time Frame: At Month 1
Population: The analysis was performed on the According-to-Protocol (ATP) cohort for immunogenicity, which included all evaluable subjects for whom immunogenicity measures were available. This primary outcome and the statistical analyses performed for this outcome concern the Nimenrix-A Group and Nimenrix-B Group only.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Nimenrix-A Group | Nimenrix-B Group | Mencevax Group
Number analyzed (Participants) | 375 | 371 | 373
Titers
  rSBA-MenA: number analyzed (Participants) | 359 | 343 | 356
  rSBA-MenA | 4846.0 [4459.8 to 5265.7] | 5064.6 [4657.5 to 5507.2] | 3421.0 [3134.7 to 3733.4]
  rSBA-MenC: number analyzed (Participants) | 374 | 370 | 372
  rSBA-MenC | 6025.4 [5269.0 to 6890.2] | 7070.7 [6225.3 to 8030.9] | 5953.1 [5188.2 to 6830.7]
  rSBA-MenW-135: number analyzed (Participants) | 375 | 370 | 372
  rSBA-MenW-135 | 9836.7 [8939.2 to 10824.3] | 8855.5 [8021.8 to 9775.9] | 4675.1 [4145.9 to 5272.0]
  rSBA-MenY | 11632.5 [10675.1 to 12675.8] | 10386.7 [9557.5 to 11287.9] | 6315.9 [5787.9 to 6892.1]
Statistical Analysis 1: Comparison: Nimenrix-A Group vs Nimenrix-B Group; Demonstration of the comparability of the immunogenicity of Lot A to Lot B of Nimenrix conjugate vaccine with respect to rSBA geometric mean titres (GMTs) for N. meningitidis serogroups A, 1 month after vaccination as measured at GSK; Test type: Non-Inferiority — Criterion for non-inferiority: Non-inferiority of Nimenrix Lot B vs. Nimenrix Lot A in terms of non-inferiority would be demonstrated if the upper limit (UL) of the 2-sided 95% CIs on the rSBA GMT ratios (GMTs of Nimenrix Lot B over the GMTs of the Nimenrix Lot A) would be below (<) a limit of 2-fold for antibodies against all meningococcal serogroups; Adjusted GMT ratio = 1.04, 95% CI 2-sided [0.92 to 1.17]
Statistical Analysis 2: Comparison: Nimenrix-A Group vs Nimenrix-B Group; Demonstration of the comparability of the immunogenicity of Lot A to Lot B of Nimenrix conjugate vaccine with respect to rSBA geometric mean titres (GMTs) for N. meningitidis serogroups C, 1 month after vaccination as measured at GSK; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; Adjusted GMT ratio = 1.15, 95% CI 2-sided [0.96 to 1.37]
Statistical Analysis 3: Comparison: Nimenrix-A Group vs Nimenrix-B Group; Demonstration of the comparability of the immunogenicity of Lot A to Lot B of Nimenrix conjugate vaccine with respect to rSBA geometric mean titres (GMTs) for N. meningitidis serogroups W-135, 1 month after vaccination as measured at GSK; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; Adjusted GMT ratio = 0.91, 95% CI 2-sided [0.8 to 1.04]
Statistical Analysis 4: Comparison: Nimenrix-A Group vs Nimenrix-B Group; Demonstration of the comparability of the immunogenicity of Lot A to Lot B of Nimenrix conjugate vaccine with respect to rSBA geometric mean titres (GMTs) for N. meningitidis serogroups Y, 1 month after vaccination as measured at GSK; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; Adjusted GMT ratio = 0.88, 95% CI 2-sided [0.78 to 0.99]

3. Secondary Outcome: Number of Subjects With rSBA-MenA, rSBA-MenC, rSBA-MenW-135 and rSBA-MenY Antibody Titers ≥ the Cut-off Value
Description: The cut-off value for the rSBA titers was greater than or equal to (≥) 1:8. The analysis was performed with the Health Protection Agency (HPA) rSBA assay.
Time Frame: At Day 0 and at Month 1
Population: The analysis was performed on the According-To-Protocol (ATP) cohort for immunogenicity, which included all evaluable subjects for whom immunogenicity measures were available. No testing was performed by the HPA assay on subjects from the Nimenrix-B Group.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix-A Group | Mencevax Group
Number analyzed (Participants) | 376 | 373
Participants
  rSBA-MenA, Day 0: number analyzed (Participants) | 366 | 368
  rSBA-MenA, Day 0 | 66 | 77
  rSBA-MenA, Month 1: number analyzed (Participants) | 376 | 372
  rSBA-MenA, Month 1 | 376 | 371
  rSBA-MenC, Day 0: number analyzed (Participants) | 367 | 368
  rSBA-MenC, Day 0 | 44 | 57
  rSBA-MenC, Month 1: number analyzed (Participants) | 375 | 372
  rSBA-MenC, Month 1 | 371 | 360
  rSBA-MenW-135, Day 0: number analyzed (Participants) | 366 | 368
  rSBA-MenW-135, Day 0 | 69 | 76
  rSBA-MenW-135, Month 1: number analyzed (Participants) | 373 | 370
  rSBA-MenW-135, Month 1 | 371 | 362
  rSBA-MenY, Day 0: number analyzed (Participants) | 364 | 367
  rSBA-MenY, Day 0 | 140 | 136
  rSBA-MenY, Month 1 | 376 | 367

4. Secondary Outcome: Number of Subjects With rSBA-MenA, rSBA-MenC, rSBA-MenW-135 and rSBA-MenY Antibody Titers ≥ the Cut-off Value
Description: The cut-off value for the rSBA titers was greater than or equal to (≥) 1:128. The analysis was performed with the Health Protection Agency (HPA) rSBA assay.
Time Frame: At Day 0 and Month 1
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix-A Group | Mencevax Group
Number analyzed (Participants) | 376 | 373
Participants
  rSBA-MenA, Day 0: number analyzed (Participants) | 366 | 368
  rSBA-MenA, Day 0 | 47 | 53
  rSBA-MenA, Month 1: number analyzed (Participants) | 376 | 372
  rSBA-MenA, Month 1 | 375 | 364
  rSBA-MenC, Day 0: number analyzed (Participants) | 367 | 368
  rSBA-MenC, Day 0 | 20 | 34
  rSBA-MenC, Month 1: number analyzed (Participants) | 375 | 372
  rSBA-MenC, Month 1 | 369 | 358
  rSBA-MenW-135, Day 0: number analyzed (Participants) | 366 | 368
  rSBA-MenW-135, Day 0 | 42 | 54
  rSBA-MenW-135, Month 1: number analyzed (Participants) | 373 | 370
  rSBA-MenW-135, Month 1 | 371 | 359
  rSBA-MenY, Day 0: number analyzed (Participants) | 364 | 367
  rSBA-MenY, Day 0 | 114 | 120
  rSBA-MenY, Month 1 | 376 | 367

5. Secondary Outcome: rSBA-MenA, rSBA-MenC, rSBA-MenW-135 and rSBA-MenY Antibody Titers
Description: Titers are presented as geometric mean titers (GMTs). The analysis was performed with the Health Protection Agency (HPA) rSBA assay.
Time Frame: At Day 0 and at Month 1
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Nimenrix-A Group | Mencevax Group
Number analyzed (Participants) | 376 | 373
Titers
  rSBA-MenA, Day 0: number analyzed (Participants) | 366 | 368
  rSBA-MenA, Day 0 | 4.7 [3.9 to 5.7] | 5.3 [4.4 to 6.5]
  rSBA-MenA, Month 1: number analyzed (Participants) | 376 | 372
  rSBA-MenA, Month 1 | 3463.4 [3152.6 to 3804.8] | 2186.0 [1923.9 to 2483.8]
  rSBA-MenC, Day 0: number analyzed (Participants) | 367 | 368
  rSBA-MenC, Day 0 | 3.2 [2.8 to 3.6] | 3.7 [3.2 to 4.4]
  rSBA-MenC, Month 1: number analyzed (Participants) | 375 | 372
  rSBA-MenC, Month 1 | 4187.9 [3563.8 to 4921.2] | 3649.1 [3026.5 to 4399.8]
  rSBA-MenW-135, Day 0: number analyzed (Participants) | 366 | 368
  rSBA-MenW-135, Day 0 | 4.8 [3.9 to 5.8] | 5.5 [4.4 to 6.8]
  rSBA-MenW-135, Month 1: number analyzed (Participants) | 373 | 370
  rSBA-MenW-135, Month 1 | 12725.1 [10998.4 to 14722.9] | 4365.4 [3622.8 to 5260.1]
  rSBA-MenY, Day 0: number analyzed (Participants) | 364 | 367
  rSBA-MenY, Day 0 | 13.3 [10.3 to 17.2] | 12.6 [9.8 to 16.3]
  rSBA-MenY, Month 1 | 5911.3 [5315.2 to 6574.3] | 2554.9 [2211.6 to 2951.4]

6. Secondary Outcome: Number of Subjects With rSBA-MenA, rSBA-MenC, rSBA-MenW-135 and rSBA-MenY Antibody Titers Above the Cut-off Value
Description: The cut-off value for the rSBA titers was greater than or equal to (≥) 1:8. The analysis was performed with the GSK rSBA assay.
Time Frame: At Day 0 and at Month 1
Population: The analysis was performed on the According-To-Protocol (ATP) cohort for immunogenicity, which included all evaluable subjects for whom immunogenicity measures were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix-A Group | Nimenrix-B Group | Mencevax Group
Number analyzed (Participants) | 375 | 371 | 373
Participants
  rSBA-MenA, Day 0: number analyzed (Participants) | 320 | 328 | 310
  rSBA-MenA, Day 0 | 296 | 314 | 295
  rSBA-MenA, Month 1: number analyzed (Participants) | 359 | 343 | 356
  rSBA-MenA, Month 1 | 359 | 343 | 356
  rSBA-MenC, Day 0: number analyzed (Participants) | 351 | 350 | 361
  rSBA-MenC, Day 0 | 211 | 213 | 224
  rSBA-MenC, Month 1: number analyzed (Participants) | 374 | 370 | 372
  rSBA-MenC, Month 1 | 374 | 370 | 372
  rSBA-MenW- 135, Day 0: number analyzed (Participants) | 343 | 333 | 345
  rSBA-MenW- 135, Day 0 | 296 | 286 | 298
  rSBA-MenW- 135, Month 1: number analyzed (Participants) | 375 | 370 | 372
  rSBA-MenW- 135, Month 1 | 375 | 370 | 372
  rSBA-MenY, Day 0: number analyzed (Participants) | 363 | 359 | 364
  rSBA-MenY, Day 0 | 335 | 338 | 336
  rSBA-MenY, Month 1 | 375 | 371 | 373

7. Secondary Outcome: rSBA-MenA, rSBA-MenC, rSBA-MenW-135 and rSBA-MenY Antibody Titers
Description: Titers are presented as geometric mean titers (GMTs). The analysis was performed with the GSK rSBA assay.
Time Frame: At Day 0
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Nimenrix-A Group | Nimenrix-B Group | Mencevax Group
Number analyzed (Participants) | 363 | 359 | 364
Titers
  rSBA-MenA: number analyzed (Participants) | 320 | 328 | 310
  rSBA-MenA | 348.4 [293.0 to 414.2] | 401.4 [347.2 to 464.1] | 424.4 [362.9 to 496.5]
  rSBA-MenC: number analyzed (Participants) | 351 | 350 | 361
  rSBA-MenC | 36.3 [29.3 to 45.0] | 44.7 [35.6 to 56.2] | 46.9 [37.2 to 59.0]
  rSBA-MenW-135: number analyzed (Participants) | 343 | 333 | 345
  rSBA-MenW-135 | 185.9 [153.1 to 225.6] | 191.2 [155.9 to 234.4] | 205.5 [167.6 to 252.0]
  rSBA-MenY | 387.5 [324.9 to 462.2] | 426.8 [362.2 to 502.8] | 412.6 [346.8 to 490.8]

8. Secondary Outcome: Number of Subjects With Vaccine Response for rSBA-MenA, rSBA-MenC, rSBA-MenW-135 and rSBA-MenY Antibodies
Description: Vaccine response defined as: for initially seronegative subjects, antibody titer greater than or equal to (≥) 1:32 and for initially seropositive subjects: antibody titer ≥ 4 fold the pre-vaccination antibody titer. The analysis was performed with the Health Protection Agency (HPA) rSBA assay.
Time Frame: At Month 1
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix-A Group | Mencevax Group
Number analyzed (Participants) | 362 | 360
Participants
  rSBA-Men | 356 | 353
  rSBA-MenC | 354 | 347
  rSBA-MenW-135: number analyzed (Participants) | 360 | 358
  rSBA-MenW-135 | 356 | 345
  rSBA-MenY: number analyzed (Participants) | 360 | 360
  rSBA-MenY | 355 | 343

9. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 pain = pain that prevented normal activity. Grade 3 redness/swelling = redness/swelling spreading beyond 50 millimeters (mm) of injection site.
Time Frame: Within 4-days (Days 0-3) post-vaccination
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects for whom data were available and who had the symptoms sheet filled in.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix-A Group | Nimenrix-B Group | Mencevax Group
Number analyzed (Participants) | 386 | 384 | 383
Participants
  Any Pain | 208 | 210 | 141
  Grade 3 Pain | 6 | 8 | 3
  Any Redness | 93 | 84 | 57
  Grade 3 Redness | 2 | 0 | 0
  Any Swelling | 57 | 63 | 42
  Grade 3 Swelling | 4 | 0 | 0

10. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms
Description: Assessed solicited general symptoms were fatigue, gastrointestinal symptoms, headache and temperature [defined as orally temperature equal to or above (≥) 37.5 degrees Celsius (°C)]. Any = occurrence of the symptom regardless of intensity grade. Grade 3 symptom = symptom that prevented normal activity. Grade 3 fever = fever higher than (>) 39.5 °C. Related = symptom assessed by the investigator as related to the vaccination.
Time Frame: Within 4-days (Days 0-3) post-vaccination
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix-A Group | Nimenrix-B Group | Mencevax Group
Number analyzed (Participants) | 386 | 384 | 383
Participants
  Any Fatigue | 117 | 110 | 115
  Grade 3 Fatigue | 1 | 3 | 0
  Related Fatigue | 113 | 100 | 109
  Any Gastrointestinal symptoms | 50 | 43 | 45
  Grade 3 Gastrointestinal symptoms | 2 | 2 | 1
  Related Gastrointestinal symptoms | 44 | 38 | 36
  Any Headache | 105 | 119 | 103
  Grade 3 Headache | 1 | 3 | 2
  Relate Headache | 96 | 111 | 95
  Any Temperature | 28 | 23 | 26
  Grade 3 Temperature | 0 | 0 | 0
  Related Temperature | 27 | 20 | 24

11. Secondary Outcome: Number of Subjects With Any Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination.
Time Frame: Within 31-days (Days 0-30) post-vaccination
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects for whom data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix-A Group | Nimenrix-B Group | Mencevax Group
Number analyzed (Participants) | 390 | 390 | 390
Participants | 103 | 94 | 86

12. Secondary Outcome: Number of Subjects With New Onset Chronic Illnesses (NOCI)
Description: NOCIs include autoimmune disorders, asthma, type I diabetes, allergies.
Time Frame: Within 31-days (Days 0-30) post-vaccination
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix-A Group | Nimenrix-B Group | Mencevax Group
Number analyzed (Participants) | 390 | 390 | 390
Participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Solicited local/general symptoms: during the 4-day post-vaccination period (Days 0-3). Unsolicited AEs: during the 31-day post-vaccination (Days 0-30). SAEs: during the entire study period (from Day 0 up to Month 1).
Arm/Group | Nimenrix-A Group | Nimenrix-B Group | Mencevax Group
All-Cause Mortality (participants affected / at risk) | 0/390 | 0/390 | 0/390
Serious Adverse Events (participants affected / at risk) | 0/390 | 1/390 | 0/390
Other Adverse Events (participants affected / at risk) | 274/390 | 271/390 | 237/390
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nimenrix-A Group (N=390) | Nimenrix-B Group (N=390) | Mencevax Group (N=390)
Blighted ovum (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Nimenrix-A Group (N=390) | Nimenrix-B Group (N=390) | Mencevax Group (N=390)
Pain (General disorders) | 208/386 | 210/384 | 141/383
Redness (General disorders) | 93/386 | 84/384 | 57/383
Swelling (General disorders) | 57/386 | 63/384 | 42/383
Fatigue (General disorders) | 117/386 | 110/384 | 115/383
Gastrointestinal (General disorders) | 50/386 | 43/384 | 45/383
Headache (General disorders) | 105/386 | 119/384 | 103/383
Temperature /(Orally) (General disorders) | 28/386 | 23/384 | 26/383

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.